CLINICAL TRIAL: NCT00178633
Title: Dramatic Reversal of Derangements in Muscle Metabolism and Left Ventricular Function After Bariatric Surgery
Brief Title: Metabolic Parameters 3 Months, 9 Months, and 2 Years After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HSC-MS-02-137; 5R01HL073162-02 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Diabetes; Heart Failure; Insulin Resistance
Keywords: Obesity; Insulin Resistance; Free Fatty Acids; Heart Failure
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Heart Failure; Insulin Resistance | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skeletal muscle biopsies, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric Surgery: Procedures were not part of the trial. Patients already undergoing these clinical procedures agreed to analysis and follow-up for research purposes. All patients had one of two different types of procedures, but outcome analyses did not distinguish between the two procedures.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery was not part of this trial. This was observational trial of persons post-bariatric surger.

SUMMARY:
An original cohort of 43 patients were recruited for analysis of anthropometrics, metabolic profile, skeletal muscle biopsy, echocardiogram at baseline, 3 months and 9 months post bariatric surgery. While all 43 patients reportedly completed 3 and 9 month evaluations, only 15 patients completed 24 month evaluations due to 28 patients unwilling to return.

The overarching purpose appears to have been not only evaluation of weightloss, but normalization of metabolic profile over time.

ELIGIBILITY:
Inclusion Criteria:

* The subjects in this study will represent both male and female patients with clinically severe obesity (BMI > 40kg/m2 or 35kg/m2 with significant obesity related co-morbidities), who have chosen to undergo elective bariatric surgery. Patients are screened through the University of Texas Houston Bariatric Surgery Center (UTHBSC) and are evaluated for bariatric surgery, defined in this study as small pouch gastric bypass with Roux-en-Y (SPGB), or laparoscopic adjustable gastric banding (LAGB). Adults (>18)from diverse ethnic backgrounds, with clinically severe obesity, are eligible to be evaluated for bariatric weight loss surgery in the UTHBSC. Candidates considered for the study are patients who not only fulfill the criteria for weight loss surgery, but also demonstrate a high likelihood of complying with the long-term follow-up that is required for a successful study.

Patients who have components of the metabolic syndrome (hypertension, diabetes, and dyslipidemia) will be included if these complications do not preclude a safe operation. .

Exclusion Criteria: Exclusion criteria include age over 70 years, current history of smoking, coronary artery disease, congestive heart failure, ischemic cardiomyopathy, known peripheral vascular disease, severe psychiatric disease, any medical problem or physical contraindication for surgery (as determined by the physician) and pregnancy. This study will be limited to adults since the safety of gastric bypass surgery has not been shown to be safe in children in large clinical trials

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female, adult patients with clinically severe obesity who have undergone elective bariatric surgery.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2004-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Taegtmeyer, MD, DPhil, Principal Investigator — University of Texas, Health Sciences Center Houston
Locations (1):
- University of Texas, Health Sciences Center Houston, Houston, Texas, United States

REFERENCES:
- [Result] Leichman JG, Aguilar D, King TM, Mehta S, Majka C, Scarborough T, Wilson EB, Taegtmeyer H. Improvements in systemic metabolism, anthropometrics, and left ventricular geometry 3 months after bariatric surgery. Surg Obes Relat Dis. 2006 Nov-Dec;2(6):592-9. doi: 10.1016/j.soard.2006.09.005. PMID 17138229
- [Result] Leichman JG, Aguilar D, King TM, Vlada A, Reyes M, Taegtmeyer H. Association of plasma free fatty acids and left ventricular diastolic function in patients with clinically severe obesity. Am J Clin Nutr. 2006 Aug;84(2):336-41. doi: 10.1093/ajcn/84.1.336. PMID 16895880
- [Result] Leichman JG, Wilson EB, Scarborough T, Aguilar D, Miller CC 3rd, Yu S, Algahim MF, Reyes M, Moody FG, Taegtmeyer H. Dramatic reversal of derangements in muscle metabolism and left ventricular function after bariatric surgery. Am J Med. 2008 Nov;121(11):966-73. doi: 10.1016/j.amjmed.2008.06.033. PMID 18954843
- [Result] Trakhtenbroit MA, Leichman JG, Algahim MF, Miller CC 3rd, Moody FG, Lux TR, Taegtmeyer H. Body weight, insulin resistance, and serum adipokine levels 2 years after 2 types of bariatric surgery. Am J Med. 2009 May;122(5):435-42. doi: 10.1016/j.amjmed.2008.10.035. PMID 19375553
- [Result] Taegtmeyer H, Leichman JG, Reyes M, Lux TR. Early benefits from weight-loss surgery. J Am Coll Cardiol. 2010 Apr 20;55(16):1754; author reply 1754. doi: 10.1016/j.jacc.2009.11.081. No abstract available. PMID 20394883
- [Result] Leichman JG, Lavis VR, Aguilar D, Wilson CR, Taegtmeyer H. The metabolic syndrome and the heart--a considered opinion. Clin Res Cardiol. 2006 Jan;95 Suppl 1:i134-41. doi: 10.1007/s00392-006-1119-7. PMID 16598541
- [Result] Taegtmeyer H, Algahim MF. Obesity and cardiac metabolism in women. JACC Cardiovasc Imaging. 2008 Jul;1(4):434-5. doi: 10.1016/j.jcmg.2008.04.008. No abstract available. PMID 19356463
- [Result] Burgmaier M, Sen S, Philip F, Wilson CR, Miller CC 3rd, Young ME, Taegtmeyer H. Metabolic adaptation follows contractile dysfunction in the heart of obese Zucker rats fed a high-fat "Western" diet. Obesity (Silver Spring). 2010 Oct;18(10):1895-901. doi: 10.1038/oby.2009.500. Epub 2010 Jan 28. PMID 20111021
- [Result] Harmancey R, Wilson CR, Wright NR, Taegtmeyer H. Western diet changes cardiac acyl-CoA composition in obese rats: a potential role for hepatic lipogenesis. J Lipid Res. 2010 Jun;51(6):1380-93. doi: 10.1194/jlr.M001230. Epub 2010 Jan 21. PMID 20093477
- [Result] Algahim MF, Lux TR, Leichman JG, Boyer AF, Miller CC 3rd, Laing ST, Wilson EB, Scarborough T, Yu S, Snyder B, Wolin-Riklin C, Kyle UG, Taegtmeyer H. Progressive regression of left ventricular hypertrophy two years after bariatric surgery. Am J Med. 2010 Jun;123(6):549-55. doi: 10.1016/j.amjmed.2009.11.020. PMID 20569762
- [Result] Ballal K, Wilson CR, Harmancey R, Taegtmeyer H. Obesogenic high fat western diet induces oxidative stress and apoptosis in rat heart. Mol Cell Biochem. 2010 Nov;344(1-2):221-30. doi: 10.1007/s11010-010-0546-y. Epub 2010 Jul 31. PMID 20676734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: IRB Approved to begin recruitment, 5.20.2004. Enrollment ended June 2006. All patients recruited from University of Texas Houston, Bariatric Surgery Center.
Period: Overall Study
Arm/Group | Bariatric Surgery
Started | 43
Completed | 37
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: 43 patients were originally enrolled, and 37 participated through 9 months; 15 female participants returned for an additional 2 year analysis.
Groups:
- Bariatric Surgery: Procedure was not part of research. Patients had already elected to undergo gastric procedure, agreed to follow up for research purposes.
Arm/Group | Bariatric Surgery
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Change in weight. Negative values represent weight loss.
Time Frame: 0 to 9 months
Population: broken out into 0-3months and 3-9months below
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Bariatric Surgery
Number analyzed (Participants) | 37
kg
  0-3 Months Post Procedure | -21.5 (18.1) [-25.0 to -18.1]
  3-9 Months Post Procedure | -16.4 [-20.1 to -12.8]
Statistical Analysis 1: Comparison: Bariatric Surgery; Test type: Superiority or Other; p < .0001, ANOVA

2. Secondary Outcome: Change in Glucose
Description: Change in glucose. Negative values represent a decrease in glucose levels.
Time Frame: 0-9 Months
Population: broken out into 0-3months and 3-9months below
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Bariatric Surgery
Number analyzed (Participants) | 37
mg/dL
  0-3 Months | -19.1 [-33.2 to -5.0]
  3-9 Months | -2.0 [-11.2 to 7.2]

3. Secondary Outcome: Change in Tissue Doppler Diastolic Velocity
Description: Change in tissue doppler diastolic velocity. Negative values indicate a decrease in tissue doppler diastolic velocity.
Time Frame: 0-9 Months
Population: Analysis broken down into 0-3 months and 3-9 months
Measure: Mean (95% Confidence Interval); unit: cm/s
Arm/Group | Bariatric Surgery
Number analyzed (Participants) | 27
cm/s
  0-3 Months | 0.4 [-.06 to 1.3]
  3-9 Months | -0.4 [-1.1 to 0.4]

4. Secondary Outcome: Change in Left Ventricular Mass
Description: Change in left ventricular mass, or myocardium, as measured in centimeters using echocardiography. Negative values represent a decrease in ventricular mass.
Time Frame: 0-9 Months
Population: broken out into 0-3months and 3-9months below
Measure: Mean (95% Confidence Interval); unit: g/m^2.7
Arm/Group | Bariatric Surgery
Number analyzed (Participants) | 37
g/m^2.7
  0-3 Month | -3.0 [-6.1 to 0.1]
  3-9 Month | -6.3 [-10.2 to -2.4]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at both 9 months and 2 years.
Groups:
- Bariatric Surgery, Follow up at 9 Months; Bariatric Surgery, Follow up at 2 Years: Procedure was not part of research. Patients had already elected to undergo gastric procedure, agreed to follow up for research purposes.
Arm/Group | Bariatric Surgery, Follow up at 9 Months | Bariatric Surgery, Follow up at 2 Years
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/19
Other Adverse Events (participants affected / at risk) | 0/37 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes